CLINICAL TRIAL: NCT00440128
Title: A Phase I, Open-Label, Randomized, Two Period Crossover Study to Investigate the Effects of GW679769 on the Pharmacokinetics of Docetaxel in Subjects With Cancer
Brief Title: The Effects Of GW679769 (Casopitant) On The Pharmacokinetics Of Docetaxel In Subjects With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NKV100781
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: Casopitant,; Neurokinin-1 Receptor Antagonist,; Drug-Interaction,; CYP3A; NK-1 Receptor Antagonist,; GW679769,; Docetaxel,
MeSH Terms: conditions — Nausea; Vomiting | interventions — Docetaxel; casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel (Active Comparator): Docetaxel
  Interventions: Drug: Docetaxel
- Docetaxel/Casopitant (Experimental): Docetaxel/Casopitant
  Interventions: Drug: Casopitant/Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel
  Arms: Docetaxel
Drug: Casopitant/Docetaxel — Casopitant/Docetaxel
  Other Names: Docetaxel; Casopitant
  Arms: Docetaxel/Casopitant

SUMMARY:
The purpose of the study is to evaluate the effect of the study drug (GW679769) on a commonly used chemotherapy drug (docetaxel) which will be given I.V. Blood samples will be taken to see if the GW679769 alters the blood levels of the chemotherapy. The study will last about 2 weeks with a final follow-up visit 6 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age
* A female is eligible to enter and participate in this study if she is of:

  1. Non-child-bearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had at least one of the following:

     * Has had a hysterectomy, or
     * Has had a bilateral oophorectomy (ovariectomy), or
     * Has had a bilateral tubal ligation, or • Is considered post-menopausal (defined as amenorrheic for ≥ 1 year) and having serum follicle stimulating hormone (FSH) and serum estradiol concentrations consistent with post-menopausal status.
  2. Childbearing potential, has a negative serum pregnancy or negative urine pregnancy test within 24 hours prior to administration of the first dose of study medication and agrees to one of the following:

     * Complete abstinence from sexual intercourse from two weeks prior to administration of the first dose of investigational product until 30 days after the final dose of study medication.
     * Use double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm) from two weeks prior to administration of the first dose of investigational product until 30 days after the final dose of study medication.
     * Vasectomized partner who has been documented to be sterile prior to the female subject's entry and is the sole sexual partner for that female.
     * NOTE: if women of childbearing potential are enrolled, they must use double-barrier contraception in addition to oral contraceptives during the active study treatment period until 6 weeks after the final dose of study medication.
* Histologically confirmed malignant solid tumor and is scheduled to receive at least 2 courses of chemotherapy with docetaxel as a single intravenous dose of 20 to 40 mg/m2 given over a duration of one hour and repeated weekly.
* Received eight or fewer previous doses of docetaxel. Subjects that have received more than eight doses of docetaxel must receive permission from the GSK medical monitor in order to be eligible for the study.
* ECOG performance status score of less than or equal to 2

NOTE: If the subject's performance status deteriorates between the screening Visit and the time of first dose of study drug to a score > 2, the subject will be excluded from the study

* Adequate hematologic and other physiological organ function as evidenced by Absolute Neutrophil Count ≥1500/mm3. Platelets ≥ 100,000/mm3 Hemoglobin ≥ 9 g/dL Serum creatinine < 1.5 mg/dL Total Bilirubin ≤ upper limit of the reference range Aspartate Transaminase (AST) < 2 x upper limit of the reference range Alanine Transaminase (ALT) < 2 x upper limit of the reference range Alkaline Phosphatase < 2.5 x upper limit of the reference range. Calculated creatinine clearance > 50 mL/min (measured by Cockcroft Gault Formula;)
* Written informed consent is obtained prior to any study-specific procedures or assessments.
* Able to swallow and retain oral medications.

Exclusion Criteria:

* Pregnant or lactating.
* Received radiation therapy to the abdomen or the pelvis in the 28 days prior to receiving the first dose of study medication or that are scheduled to receive radiation therapy to the abdomen or the pelvis in the six days following the first dose of study medication.
* Received a dose of docetaxel during the week prior to Day -1.
* Known central nervous system primary or metastatic malignancy, unless successfully treated with excision or radiation and has been stable for at least 3 months prior to receiving the first dose of study medication.
* Active systemic infection or any poorly controlled medical condition (other than malignancy) which, in the opinion of the investigator, may confound the results of the study or pose an unwarranted risk to the subject. Subjects with a previous, but not current, history of alcoholism may be permitted provided that, in the investigator's opinion, the subject's disease state will not confound the results of the study.
* Receiving regular treatment with high dose systemic corticosteroid therapy or steroid dose within 72 hours prior to receiving the first dose of study medication. Topical steroids and inhaled corticosteroids with a steroid dose of less than or equal to 10 mg prednisone daily (or its equivalent) are permitted if the subject has been on this dose for at least 14 days prior to dosing.
* Hypersensitivity or contraindication to ondansetron or other 5-HT3 receptor antagonist, dexamethasone, docetaxel, casopitant, or any component of the above mentioned medications.
* Received an investigational drug within the 28 days or five half-lives (whichever is longer) prior to receiving the first dose of study medication, or is scheduled to receive any investigational drug during the study.
* Use of strong inhibitors of CYP3A4 or CYP3A5 prior to the first dose of study medication
* Use of inducers of CYP3A4 or CYP3A5 (other than steroids described in Exclusion Criteria 5) within 14 days prior to the first dose of study medication
* Use of drugs with a narrow therapeutic index that interact with the P-glycoprotein pathway within 14 days prior to the first dose of study medication until 14 days after the last dose of docetaxel including digoxin.
* Use of drugs with a narrow therapeutic index that are metabolized by CYP2C8 within 14 days prior to the first dose of study medication including repaglinide and torsemide.
* Disease that will significantly affect absorption of oral medications.
* Inadequate venous access for pharmacokinetic sampling.
* Unresolved Grade 2 or worse toxicity from prior therapy.
* Active peptic ulcer disease (PUD) or a history of PUD of unknown etiology. NOTE: Subject is eligible to enter and participate in this study if they have a history of PUD of known etiology with documentation from a gastroenterologist or other qualified physician of the etiology of the PUD and that effective treatment was provided with full eradication of ulcers and symptoms. Subjects who present with symptoms of gastroesophageal reflux disease (GERD) are eligible. However, if the investigator suspects PUD in such a subject, the subject must have a GI assessment to rule out PUD. If assessment is negative, subject may enter the study. For these subjects, appropriate steps must also have been taken to minimize the risk of reoccurrence. If PUD was non-steroidal anti-inflammatory drug (NSAID) induced, the subject should no longer be taking NSAID medication(s). If PUD was induced by H. pylori, the subject should have been appropriately treated.
* Stool positive for occult blood. Test may be repeated once if subject did not abstain from red meat for the previous three days.
* Pepsinogen level below the lower limit of laboratory reference range (LLRR).
* Troponin level above 10% of the coefficient of variation of the assay as determined by the laboratory performing the test.
* Calculated QT interval (QTc) > 480 msecs.
* Clinically significant cardiac disease that would interfere with participation in the study as determined by the investigator.
* Known or suspected iron deficiency.
* Use of NSAIDS, including aspirin at any dose, and including COX2 inhibitors. These medications are prohibited 7 days prior to administration of study drug and for the duration of the study until 72 hours after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05-04 (Actual); Primary Completion 2008-07-17 (Actual); Study Completion 2008-07-17 (Actual)

PRIMARY OUTCOMES:
Plasma levels of study drugs will be taken on Day 1 & 8. | taken on Day 1 & 8.
  Plasma samples of study drugs

SECONDARY OUTCOMES:
Safety is evaluated by: -AEs monitored at each visit | starting at Day 1.
-Physical exam, vital signs, & ECOG performance status score | at Screening, Day 1,8,&15.
-ECG | at Screening & Day 15.
-Serum Pepsinogen levels monitored | at Screening & Followup
Terminal half-life (t1/2, as data permit), AUC(0-t), volume of distribution at steady state (Vdss), and clearance (Cl) of docetaxel | on Day 1 and 8.
Lowest measured absolute neutrophil count. | on Day 1 and 8
Physical exam findings, blood pressure, heart rate, clinical laboratory tests, clinical monitoring/observation, and adverse events reporting. | on Day 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dandamudi UB, Adams LM, Johnson B, Bauman J, Morris S, Murray S, Webb RT, Gartner E, Hohl R, Lewis LD. Lack of effect of casopitant on the pharmacokinetics of docetaxel in patients with cancer. Cancer Chemother Pharmacol. 2011 Apr;67(4):783-90. doi: 10.1007/s00280-010-1381-2. Epub 2010 Jun 17. PMID 20556613
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study NKV100781 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NKV100781?search=study&study_ids=NKV100781#rs
- Available data/document: Statistical Analysis Plan: NKV100781 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKV100781 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKV100781 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKV100781 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKV100781 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKV100781 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKV100781 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register